CLINICAL TRIAL: NCT00002355
Title: A Randomized Comparison of Immediate Versus Delayed Treatment With Intravitreal Injections of ISIS 2922 in Patients With Peripheral Cytomegalovirus (CMV) Retinitis
Brief Title: A Comparison of ISIS 2922 Used Immediately or Later in Patients With Cytomegalovirus (CMV) of the Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 251A; ISIS 2922-CS2
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents; Cytomegalovirus Retinitis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — fomivirsen

INTERVENTIONS:
Drug: Fomivirsen sodium

SUMMARY:
To determine a clinically safe and effective dose of intravitreally injected ISIS 2922 and to compare the safety and efficacy of immediate versus delayed treatment in AIDS patients with previously untreated, peripheral cytomegalovirus ( CMV ) retinitis.

DETAILED DESCRIPTION:
In Stage 1 (dose escalation), patients receive either 75 or 150 mcg intravitreal ISIS 2922. In Stage 2 (randomization), patients are enrolled in either the immediate treatment group or delayed treatment group. Immediate treatment consists of intravitreal ISIS 2922 every 7 days for 3 injections (Induction) then every 14 days for 18 weeks (Maintenance). Patients in the delayed treatment group receive no immediate anti-CMV treatment but are monitored weekly for disease progression. If disease progresses, patient receives ISIS 2922 on an identical dosage regimen as those on immediate treatment. Patients may continue ISIS 2922 on a biweekly extended maintenance schedule if dose is considered safe and the CMV retinitis is clinically controlled. Per 2/8/96 amendment, patients are now in Stage 2 at 150 mcg.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS.
* Clinical diagnosis of previously untreated peripheral CMV retinitis in one eye.
* Leading edge of a CMV retinitis lesion is at least 750 microns from zone one. NOTE:
* Patients with CMV retinitis in zone three only may be eligible if the lesions can be reliably photographed to follow progression.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions in the eye to be treated are excluded:

* External ocular infections.
* Other herpetic infections of the retina, toxoplasma retinochoroiditis, or other disease of the fundus.
* Ocular conditions that will obstruct visualization of the posterior ocular structures.
* Retinal detachment.
* Silicone oil in eye.

Patients with the following other symptoms or conditions are excluded:

* Known or suspected allergy to phosphorothioate oligonucleotides.
* Syphilis.
* Pseudoretinitis pigmentosa.

Concurrent Medication:

Excluded:

* Current treatment for extra-ocular CMV infection.
* Ganciclovir.
* Foscarnet.
* Mellaril.
* Stelazine.
* Thorazine.
* Clofazimine.
* Ethambutol/fluconazole combination.
* Investigational medications for CMV retinitis.

Concurrent Treatment:

Excluded:

* Investigational procedures for CMV retinitis.

Patients with the following prior conditions are excluded:

* History of surgery to correct retinal detachment in the eye to be treated.
* History of syphilis.

Prior Medication:

Excluded:

* Prior anti-CMV retinitis treatment in either eye.
* Anti-CMV therapy for extra-ocular infection within the past 2 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Retina - Vitreous Associates Med Group, Los Angeles, California
  - Community Eye Med Group, Pasadena, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Dr Julio Perez, Fort Lauderdale, Florida
  - Georgia Retina, Atlanta, Georgia
  - Univ of Illinois, Chicago, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - Vitreo - Retinal Consultants, New York, New York
  - Charlotte Eye Ear Nose & Throat Association, Charlotte, North Carolina
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Novum Inc, Seattle, Washington